CLINICAL TRIAL: NCT06745544
Title: Impact of Screening and Multicomponent Exercise on Fall Rates, Fractures, and Cardiovascular Health in Diabetes: Protocol for a Randomized Control Trial: DIACTIVE
Brief Title: Impact of Screening and Multicomponent Exercise on Fall Rates, Fractures, and Cardiovascular Health in Diabetes
Acronym: DiaACTIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other); Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Nicklas Højgaard-hessellund Rasmussen, Associate Professor, MD, PhD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N-20240025; NNF22SA0079901 (Other Grant/Funding Number: the Danish Diabetes and Endocrine Academy, which is funded by the Novo Nordisk Foundation)
Record Dates: First submitted 2024-11-28; First posted 2024-12-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes; Osteoporosis; Diabetic Neuropathies; Fall Prevention; Cardiovascular Diseases
Keywords: Diabetes; T1D; T2D; RYMA; Falls; Neuropathy; CVD; Diabetic Complications; Bone health; Fractures
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Osteoporosis; Diabetic Neuropathies; Cardiovascular Diseases; Diabetes Mellitus; Diabetes Complications; Fractures, Bone | interventions — Activities of Daily Living; Exercise

STUDY DESIGN:
Intervention Model Description: The study follows a randomized controlled trial design. Participants are randomly allocated to either the 26 weeks RYMA/ADL exercise intervention group or the control group (usual care). Baseline measures are performed at day 0. Then, follow-up regardless of group is after 26, 52 and 104 weeks and a final visit after 5 years from baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- RYMA group (Experimental): Participants in this arm will engage in the Rhythm- and Multitask-Based Activity (RYMA) exercise program, a multicomponent intervention that combines strength, balance, coordination, and cognitive-motor training. The intervention also incorporates Activities of Daily Living (ADL)-based exercises to address real-world functional needs. The program is delivered over 26 weeks and includes music-based exercises designed to improve fall prevention, bone health, and cardiovascular outcomes.
  Interventions: Other: Rhythm- and Multitask-Based Activity (RYMA) and Activities of Daily Living (ADL)
- Usual Care/No Structured Exercise Intervention (No Intervention): Participants in this arm will continue their usual daily routines without any structured exercise intervention during the first 26 weeks.
- Control Group without diabetes (No Intervention): Healthy controls without diabetes equally divided between men and women without diabetes for baseline comparisons.

INTERVENTIONS:
Other: Rhythm- and Multitask-Based Activity (RYMA) and Activities of Daily Living (ADL) — The Rhythm- and Multitask-Based Activity (RYMA) program is a unique cognitive-motor exercise intervention designed for older adults with diabetes. It incorporates rhythm-based multitasking exercises, performed to improvised piano music, combined with Activities of Daily Living (ADL)-focused exercises. The intervention targets physical (strength, balance, and coordination) and cognitive (executive function, reaction time) components to reduce fall risk, improve bone health, and optimize cardiovascular outcomes. Delivered over 26 weeks, the program emphasizes social interaction to enhance adherence and long-term engagement.
  Other Names: Exercise; training; balance training
  Arms: RYMA group

SUMMARY:
The DIACTIVE study is a randomized controlled trial with a 5- year follow-up designed to evaluate the impact of comprehensive screening and multicomponent interventions on fall prevention, bone health, nerve function and cardiovascular outcomes in people with diabetes aged 65 years and older on the short and longer term. Diabetes significantly increases risks of falls, fractures, and cardiovascular disease, yet these areas remain underexplored in clinical research. This trial addresses these gaps with a novel, multidimensional approach.

Participants undergo extensive baseline assessments, including fall risk stratification, bone mineral density measurements via DXA scans, neuropathy evaluations, and cardiovascular profiling. Based on these evaluations, participants are allocated to risk-based intervention arms. The study's centerpiece is the RYMA and ADL exercise program, a tailored cognitive-motor training regimen integrating strength, balance, and executive function exercises with music-based coordination tasks. Pharmacological treatments for osteoporosis and optimization of cardiovascular risk profiles (e.g., SGLT2 inhibitors, GLP-1 agonists) are also incorporated.

Primary outcomes focus on reducing fall rates by at least 30%, improving bone density, mitigating fracture risks, enhancing nerve function, and lowering cardiovascular event rates. Secondary endpoints explore mechanisms underlying fall reduction, quality of life improvements, and adherence to interventions. Advanced methodologies such as gait analysis, seismocardiography, and magnetic resonance imaging (MRI) provide detailed insights into the intervention's effects. Follow-ups at 26 weeks, 52 weeks, 2 years, and 5 years ensure long-term efficacy evaluation.

This trial is conducted at Steno Diabetes Center North and involves interdisciplinary collaboration. By addressing key complications of diabetes through integrated care, the study aims to improve patient outcomes and inform future healthcare strategies for older people with diabetes.

DETAILED DESCRIPTION:
The DIACTIVE study is a randomized controlled trial with a 5-year follow-up designed to assess the effectiveness of a comprehensive intervention targeting fall prevention, bone health, nerve function and cardiovascular outcomes in people with diabetes aged 65 years and older. This innovative research seeks to address critical health vulnerabilities associated with diabetes, particularly the elevated risks of falls, fractures, and cardiovascular diseases (CVD). The study's integrated approach involves advanced screening techniques, tailored interventions, and long-term follow-ups, providing new insights into diabetes management for older populations. Diabetes mellitus (DM) is a chronic condition with rising global prevalence, projected to affect over 783 million people by 2045. While much attention has been given to micro- and macrovascular complications, less focus has been placed on other significant diabetes-related concerns such as bone health, neuropathy, and fall risk. Diabetes exacerbates age-related declines in musculoskeletal strength, sensory function, and cardiovascular resilience, increasing risks of falls and fractures. The interplay between these factors remains underexplored, necessitating multidimensional approaches to care. The DIACTIVE trial addresses these gaps by integrating advanced fall screening, comprehensive bone health evaluations, and cardiovascular profiling with targeted interventions. Its cornerstone is the RYMA exercise program, a novel, music-based training regimen that combines physical and cognitive elements to enhance balance, strength, and executive function.

The study has several primary objectives: reducing fall rates by 30% after 26 weeks of intervention, sustained at 52 weeks and beyond; improving bone mineral density (BMD) and mitigating fracture risks; lowering cardiovascular event rates and improving key cardiovascular markers; enhancing nerve function and reducing the progression of diabetic peripheral neuropathy (DPN); and improving psychological and social outcomes, including reduced fear of falling, enhanced mobility, and better mental well-being. This trial adopts a prospective, randomized controlled design and includes recruitment and screening of people aged ≥65 years with T1D or T2D from outpatient diabetes clinics. Participants undergo comprehensive baseline assessments, including DXA scans for BMD, fall risk stratification, neuropathy evaluations, and cardiovascular profiling using blood pressure, ECG, and advanced imaging techniques like MRI and seismocardiography. Based on their risk profiles, participants are randomized into intervention and control groups. The intervention group engages in the RYMA exercise program, which combines physical and cognitive training elements, including multitasking, reaction-based exercises, and coordination tasks, set to improvised piano music. Pharmacological treatments for osteoporosis and cardiovascular optimization are implemented as per ADA and local guidelines. Outcomes are assessed at 26 weeks, 52 weeks, 2 years, and 5 years, covering fall rates, BMD, nerve function, cardiovascular health, and quality of life.

The RYMA exercise program is the core intervention and focuses on cognitive-motor training through rhythm-based exercises. It targets key risk factors for falls by improving balance, strength, executive function, and coordination while integrating social elements to enhance adherence and sustainability. Bone health interventions involve stratification based on DXA results, with pharmacological treatments for osteoporosis provided according to ADA guidelines. Cardiovascular optimization includes medications such as SGLT2 inhibitors, GLP-1 receptor agonists, and statins, tailored to the participants' risk profiles. The study's primary endpoints include reducing fall rates, improving BMD, reducing fracture risk, optimizing cardiovascular outcomes, and enhancing nerve function. Secondary endpoints focus on understanding the mechanisms underlying these improvements, quality-of-life metrics, and participant adherence to the interventions.

Assessments include validated fall risk algorithms, DXA scans, neuropathy tests (e.g., NC-Stat DPNCheck, vibration perception thresholds, and sensory testing), cardiovascular imaging (e.g., MRI, seismocardiography), and cognitive and physical performance evaluations. Gait analysis, postural stability, muscle strength, and executive function tests provide insights into the intervention's mechanistic effects. The trial aims to recruit 440 participants (220 T1D and 220 T2D). Inclusion criteria are: age ≥65 years, confirmed diagnosis of diabetes for at least one year, and the ability to live independently and participate in the exercise program. Exclusion criteria include severe cognitive impairment, neurological or orthopedic conditions affecting mobility, and participation in other interventional studies within six months.

This study represents a paradigm shift in diabetes management by addressing interconnected health risks through a holistic approach. Its multidisciplinary interventions combine physical, cognitive, and pharmacological elements to improve outcomes in older people with diabetes. By targeting fall prevention, bone health, and cardiovascular risk factors simultaneously, DIACTIVE has the potential to significantly enhance the quality of life and inform future healthcare strategies. Findings from the study will contribute to clinical guidelines, emphasizing integrated care models and tailored interventions for high-risk populations. Long-term follow-ups will provide critical data on the sustainability and scalability of such programs, paving the way for broader implementation in healthcare systems

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with either T1D or T2D with a minimum of 65 years of age with no upper limit.
2. Living in their own home
3. A diagnosis of diabetes at least one year prior to inclusion of the study to avoid honeymoon diabetes.
4. Signed the informed consent.

Exclusion Criteria:

1. No previous experience with rhythm-based multitask exercise.
2. Having significant neurological diseases (e.g., Parkinson's and Multiple Sclerosis), vestibular diseases, or orthopedic surgeries (e.g., hip/knee replacement) affecting their ability to participate in the study.
3. Having severely impaired cognitive function, defined as a score below 8 on the cognitive assessment "the short orientation-memory-concentration test."
4. Being fully dependent on walking aids.
5. Pregnancy or breast feeding
6. Active malignancy or terminally ill.
7. Not being able to understand Danish written and/or verbally.
8. Participating in other interventional clinical studies within the last six months
9. People with a weekly exercise activity above 5 hours a week

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Male and females
Enrollment: 490 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in Fall Rates | Measurements will take place at 26 weeks, 52 weeks, 104 weeks, and 5 years post-intervention to evaluate both short- and long-term effects of the intervention.
  To estimate changes in fall rates in people with T1D and T2D diabetes aged >65 after RYMA intervention. Fall rates will be compared to participants' baseline measures (self-controls) and to a usual care group (no RYMA).
Improvement in Bone Mineral Density (BMD) | Measurements will assess changes at 26 weeks, 52 weeks, 104 weeks, and 5 years post-intervention to evaluate sustained benefits.
  The primary outcome is to measure change in bone mineral density (BMD) after 26 weeks of intervention compared to baseline and the control group. BMD will be assessed using dual-energy X-ray absorptiometry (DXA) scans at key anatomical sites, including the lumbar spine and femoral neck. Fracture incidence will also be tracked during the follow-up period
Reduction in Cardiovascular Risk and Events | 26 weeks, 52 weeks, 104 weeks, and 5 years post-intervention.
  To estimate the change of cardiovascular risk factors on microvascular and cardiac function in people at high risk for CVD when intervented with RYMA intervention. This will be assessed using high-frequency echocardiography for detailed imaging of the heart and aorta, and magnetic resonance imaging (MRI) to evaluate cardiac structure and function.
Improvement in Nerve Function | 26 weeks, 52 weeks, 104 weeks, and 5 years post-intervention.
  To estimate the change of nerve fiber function by determining the degree of small, large and autonomic neuropathy after RYMA and cardiovascular optimization.
Blood glucose changes | HbA1c measurements will take place at baseline and after 26 weeks, 52 weeks, 104 weeks, and 5 years post-intervention to evaluate both short- and long-term effects of the intervention. CGM will be measures blinded during the 26 weeks RYMA intervention.
  To estimate changes in blood glucose levels in people with T1D and T2D diabetes aged >65 after RYMA intervention. Measures includes HbA1c and blinded continuous Glucose monitoring (CGM). Glucose levels will be compared to participants' baseline measures (self-controls) and to a usual care group (no RYMA). CGM measures will take place during the RYMA intervention

SECONDARY OUTCOMES:
Mechanisms associated with Fall Reduction | 26 weeks, 52 weeks, 104 weeks, and 5 years post-intervention
  Secondary outcomes include investigating the mechanisms underlying fall reduction. These will be assessed through gait analysis, postural stability tests, and muscle strength evaluations (e.g., handgrip strength and knee extension). Changes in cognitive function, particularly executive functions like decision-making and reaction time, will also be measured. The outcomes aim to provide insights into how the intervention impacts fall risk factors
Improvement in Quality of Life | 26 weeks, 52 weeks, 104 weeks, and 5 years post-intervention
  Secondary outcomes include changes in quality of life as measured by validated instruments such as the EQ-5D and Falls Efficacy Scale. These assessments will evaluate physical, emotional, and social well-being, including reduced fear of falling and increased confidence in performing daily activities. Changes will be tracked longitudinally.
Reduction in Fracture Risk | 52 weeks, 104 weeks, and 5 years post-intervention.
  Secondary outcomes include a changes in fracture incidences over the study period. Fractures will be recorded through participant reports and verified via medical records. Risk reduction will be analyzed in relation to improvements in bone mineral density and fall rates.
Improvement in Cardiovascular Function | 26 weeks, 52 weeks, 104 weeks, and 5 years post-intervention.
  Secondary outcomes include changes in cardiovascular function, assessed through imaging techniques such as cardiac MRI and seismocardiography, as well as biochemical markers like NT-proBNP and hs-CRP. Functional capacity will also be evaluated through tests like the 6-minute walk test.
Improvement in Cognitive Function | 26 weeks, 52 weeks, 104 weeks, and 5 years post-intervention.
  Secondary outcomes include changes in cognitive function, particularly in executive functions such as attention, memory, and problem-solving. These will be assessed using validated neuropsychological tests and reaction time measures.
Membran properties | year 2 and year 5
  To evaluate changes in nerve membrane properties including shifts in ion-channel composition or activity.

OTHER OUTCOMES:
Sustainability of Intervention Effects | 2 years and 5 years post-intervention.
  Exploratory outcomes include the sustainability of changes in fall rates, bone health, cardiovascular markers, and neuropathy beyond the primary study follow-up period. This will assess whether the intervention's effects persist after the active program ends, particularly focusing on fall prevention and quality-of-life metrics.
Changes in Muscle Mass and Composition | 26 weeks, 52 weeks, 104 weeks, and 5 years post-intervention.
  Exploratory outcomes include changes in muscle mass and body composition as measured by DXA scans. These outcomes will evaluate whether the intervention influences muscle quality, fat distribution, and sarcopenia risk over time, with comparisons between intervention and control groups
Changes in Inflammatory Biomarkers | 26 weeks, 52 weeks, and 104 weeks post-intervention.
  Exploratory outcomes include changes in systemic inflammation, assessed through biomarkers. These outcomes aim to evaluate potential mechanisms linking reduced inflammation to improved cardiovascular and bone hea

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center North, Aalborg, Norh, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data related to primary and secondary outcomes will be shared. This includes data on fall rates, bone mineral density, neuropathy, cardiovascular markers, and quality of life assessments. The data will exclude any personally identifiable information and will be shared in compliance with ethical guidelines and data privacy regulations and upon reasonable request from qualified researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: It will be made available one year after the study period ends including the following year.
Access Criteria: Access to the IPD and supporting information will be granted to qualified researchers who submit a formal request and provide a detailed research proposal outlining the intended use of the data. Requests will be reviewed by the study team or a designated oversight committee to ensure appropriate use. Approved researchers will receive de-identified data and supporting documentation, such as the study protocol, statistical analysis plan, and informed consent forms, through a secure online repository.
URL: https://stenodiabetescenter.rn.dk/

REFERENCES:
- [Background] Rolke R, Magerl W, Campbell KA, Schalber C, Caspari S, Birklein F, Treede RD. Quantitative sensory testing: a comprehensive protocol for clinical trials. Eur J Pain. 2006 Jan;10(1):77-88. doi: 10.1016/j.ejpain.2005.02.003. PMID 16291301
- [Background] Mahalingasivam AA, Jespersen AK, Ejskjaer N, Hougaard DD, Vestergaard P, Rasmussen NH, Roikjer J. The co-existence of peripheral and vestibular neuropathy in diabetes: a cross-sectional study. Eur Arch Otorhinolaryngol. 2024 Feb;281(2):663-672. doi: 10.1007/s00405-023-08130-6. Epub 2023 Jul 29. PMID 37515636
- [Background] Jansen S, Bhangu J, de Rooij S, Daams J, Kenny RA, van der Velde N. The Association of Cardiovascular Disorders and Falls: A Systematic Review. J Am Med Dir Assoc. 2016 Mar 1;17(3):193-9. doi: 10.1016/j.jamda.2015.08.022. Epub 2015 Oct 9. PMID 26455926
- [Background] Rajbhandari J, Fernandez CJ, Agarwal M, Yeap BXY, Pappachan JM. Diabetic heart disease: A clinical update. World J Diabetes. 2021 Apr 15;12(4):383-406. doi: 10.4239/wjd.v12.i4.383. PMID 33889286
- [Background] Kressig RW, Allali G, Beauchet O. Long-term practice of Jaques-Dalcroze eurhythmics prevents age-related increase of gait variability under a dual task. J Am Geriatr Soc. 2005 Apr;53(4):728-9. doi: 10.1111/j.1532-5415.2005.53228_2.x. No abstract available. PMID 15817027
- [Background] Lord SR, Close JCT. New horizons in falls prevention. Age Ageing. 2018 Jul 1;47(4):492-498. doi: 10.1093/ageing/afy059. PMID 29697780
- [Background] Wollesen B, Wildbredt A, van Schooten KS, Lim ML, Delbaere K. The effects of cognitive-motor training interventions on executive functions in older people: a systematic review and meta-analysis. Eur Rev Aging Phys Act. 2020 Jul 2;17:9. doi: 10.1186/s11556-020-00240-y. eCollection 2020. PMID 32636957
- [Background] Sherrington C, Fairhall N, Kwok W, Wallbank G, Tiedemann A, Michaleff ZA, Ng CACM, Bauman A. Evidence on physical activity and falls prevention for people aged 65+ years: systematic review to inform the WHO guidelines on physical activity and sedentary behaviour. Int J Behav Nutr Phys Act. 2020 Nov 26;17(1):144. doi: 10.1186/s12966-020-01041-3. PMID 33239019
- [Background] Rasmussen NH, Dal J, den Bergh JV, de Vries F, Jensen MH, Vestergaard P. Increased Risk of Falls, Fall-related Injuries and Fractures in People with Type 1 and Type 2 Diabetes - A Nationwide Cohort Study. Curr Drug Saf. 2021;16(1):52-61. doi: 10.2174/1574886315666200908110058. PMID 32900349
- [Background] Langdahl BL, Hofbauer LC, Forfar JC. Cardiovascular Safety and Sclerostin Inhibition. J Clin Endocrinol Metab. 2021 Jun 16;106(7):1845-1853. doi: 10.1210/clinem/dgab193. PMID 33755157
- [Background] Rasmussen NH, Dal J. Falls and Fractures in Diabetes-More than Bone Fragility. Curr Osteoporos Rep. 2019 Jun;17(3):147-156. doi: 10.1007/s11914-019-00513-1. PMID 30915638
- See also: Related Info — https://stenodiabetescenter.rn.dk/